CLINICAL TRIAL: NCT07123922
Title: Effect of Silymarin as Add on Therapy on Oxidative Stress, Pulmonary Function and Quality of Life in Stable COPD Patients; A Randomized Double-Blind Placebo-Controlled Trial
Brief Title: Effect of Silymarin as Add on Therapy on Oxidative Stress, Pulmonary Function and Quality of Life in Stable COPD Patients.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Sanjida Akter, Sanjida Akter, MD, Bangabandhu Sheikh Mujib Medical University, Dhaka., Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BSMMU/2025/4267
Record Dates: First submitted 2025-06-18; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Silymarin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silymarin (Experimental): Participants received Cap. Silymarin 140 mg orally thrice daily for 12 weeks
  Interventions: Dietary Supplement: Silymarin
- Placebo (Placebo Comparator): Participants received Silymarin placebo capsule matching Silymarin orally thrice daily for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Silymarin — Participants received Silymarin 140 mg capsule orally thrice daily for 12 weeks
  Arms: Silymarin
Dietary Supplement: Placebo — Participants received Silymarin placebo capsule thrice daily for 12 weeks
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if Silymarin works to reduce oxidative stress, improve pulmoary function and quality of life in stable COPD patients. It will also learn about the safety of drug Silymarin. The main questions it aims to answer are:

Does drug Silymarin reduce oxidative stress, improve pulmonary function and quality of life in stable COPD patients? What medical problems do participants have when taking drug Silymarin? Researchers will compare Silymarin to a placebo (a look-alike substance that contains no drug) to see if Silymarin works to treat COPD.

Participants will:

Take Silymarin or a placebo thrice daily every day for 3 months. Baseline and 3 months after plasma Malondealdehyde, erythrocyte Glutathione , FEV1, SGRQ-C score will be monitored.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a leading cause of morbidity and mortality worldwide, characterized by persistent airflow limitation and an exaggerated inflammatory response. Oxidative stress plays a pivotal role in disease progression, contributing to worsening pulmonary function, increased exacerbations, and poor quality of life. Current pharmacological interventions, including inhaled corticosteroids (ICS), bronchodilators, and mucolytics (e.g., acetylcysteine, carbocysteine, erdosteine), have limitations such as increased risk of infections, systemic side effects, and suboptimal long-term efficacy in mitigating oxidative stress. Antioxidant vitamins (A, C, E) have been explored for oxidative stress management but demonstrate inconsistent clinical benefits.

Silymarin, a bioflavonoid complex derived from Silybum marianum, possesses potent antioxidant, anti-inflammatory, and hepatoprotective properties. Silymarin is safe in human at therapeutic doses and is well tolerated even at high dose of 700 mg three times a day for 24 weeks. It scavenges reactive oxygen species (ROS), upregulates endogenous antioxidant defense mechanisms, and modulates inflammatory pathways, making it a promising candidate for managing oxidative stress in COPD. Despite extensive use in hepatic disorders, its therapeutic potential in pulmonary diseases remains underexplored.

Aim: This study aims to evaluate the effect of Silymarin on oxidative stress, pulmonary function, and quality of life in stable COPD patients.

Methodology: This research will be conducted in Pharmacology department of Bangabandhu Sheikh Mujib Medical University (BSMMU) and outpatient department of Respiratory Medicine of BSMMU from the day of approval by IRB to January, 2026. It will be single centered, randomized, double-blind, placebo-controlled trial involving stable COPD patients receiving 'Indacaterol plus Glycopyrronium'. 70 Participants will be enrolled, 35 in each group, randomly assigned to receive either Silymarin 140 mg thrice daily or placebo thrice daily for 12 weeks period. The primary outcome will be changes in oxidative stress markers (e.g., malondialdehyde, erythrocyte glutathione). Secondary outcomes include pulmonary function test (FEV1), quality of life (SGRQ-C scores). Data will be collected about various socio-demographic variables such as age, sex, smoking history, other co-morbidities. Silymarin 140 mg capsule and placebo will be purchased from Square Pharmaceutical Limited. We have an initial discussion and have a commitment that they will provide medicine and placebo along with quality control certificate. Descriptive statistics will be used for demographic variables. Means and standard deviation for continuous variables and number, percentage for categorical variables will be used. For independent samples; t-test will be utilized to analyze the average differences in MDA conc., erythrocyte glutathione conc. between the group receiving Silymarin supplement and the group receiving placebo. The Chi-square test will be employed to compare the percentage of participants may show a significant change in MDA, erythrocyte glutathione conc. in the group that received Silymarin versus the group that received placebo. Pearson or Spearman correlation tests will be used to explore any relationships between baseline MDA, erythrocyte glutathione conc. and baseline FEV1, SGRQ-C score as well as change among in MDA, erythrocyte glutathione conc. and the change in FEV1, SGRQ-C score. This study will adhere to ethical guidelines for human research, ensuring informed consent, patient safety, and data confidentiality.

Conclusion: Given the limitations of current antioxidant therapies in COPD, Silymarin offers a novel, potentially safer approach to mitigating oxidative stress and improving patient outcomes. If effective, it could serve as an adjunctive therapy to conventional COPD management, reducing the reliance on ICS and mucolytics while addressing the underlying pathophysiology of the disease and mitigating disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed case of COPD according to GOLD guideline (post bronchodilator FEV1/FVC < 0.7).
* Age 40-80 years
* No exacerbation or hospitalization due to exacerbation in the last 1 month.

Exclusion Criteria:

* • COPD exacerbation

  * Presence of other respiratory diseases like asthma, bronchiectasis, interstitial lung disease, tuberculosis or lung cancer
  * Diagnosed case of diabetes mellitus, liver disease, heart disease, kidney stones and disease, hyperparathyroidism, other malignancies
  * Use of other antioxidant drugs like Vitamin C, E, N acetylcysteine within last 1 months
  * Known hypersensitivity to Silymarin

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Oxidative stress marker plasma MDA | 12 weeks
  Comparison of plasma malondialdehyde (MDA) between control and intervention arms at baseline and after 12 weeks of treatment.
Oxidative stress marker erythrocyte glutathione | 12 weeks
  Comparison of erythrocyte glutathione concentration (GSH) between control and intervention arms at baseline and after 12 weeks of treatment.

SECONDARY OUTCOMES:
Pulmonary function | 12 weeks
  Comparison of forced expiratory volume in first second (FEV1) in Spirometry between control and intervention arms at baseline and after 12 weeks of treatment.
SGRQ-C score | 12 weeks
  Comparison of score of St. George's Respiratory Questionnaire (SGRQ-C) between control and intervention arms at baseline and after 12 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- BSMMU, Dhaka, Bangladesh